CLINICAL TRIAL: NCT00237861
Title: Effectiveness of Atypical Vs Conventional Antipsychotics
Brief Title: Effectiveness of Atypical Versus Conventional Antipsychotics in Treating Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH57292; R01MH057292 (NIH)
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Olanzapine; Quetiapine Fumarate

INTERVENTIONS:
Drug: risperidone
Drug: olanzapine
Drug: quetiapine

SUMMARY:
This study will compare the effectiveness of newer atypical antipsychotics versus older conventional antipsychotics in treating schizophrenia.

DETAILED DESCRIPTION:
At seven participating hospitals, acutely exacerbated patients with schizophrenia were randomly assigned to treatment with antipsychotic from the atypical class vs antipsychotic from the conventional class. Medication choice within class, dose, concomitant medications, and other prescribing decisions were left to the community prescriber. Patients were followed for one year after discharge.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized for schizophrenia

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
PANSS
Retention.

SECONDARY OUTCOMES:
EPS, TD.

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Woods, MD, Principal Investigator — Yale University